CLINICAL TRIAL: NCT00229996
Title: Oral Contraceptives Versus Depot-Leuprolide Taken After Surgery for Endometriosis-Associated Pelvic Pain
Brief Title: Medical Treatment of Endometriosis-Associated Pelvic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01HD044870 (NIH)
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Endometriosis; Pelvic Pain
Keywords: endometriosis; pelvic pain; treatment
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Contraceptives, Oral; Norethindrone

INTERVENTIONS:
Drug: Oral Contraceptive
Drug: Depot-Leuprolide/Norethindrone

SUMMARY:
The Specific Aim of this project is to compare the efficacy and cost-effectiveness of continuous oral contraceptives versus leuprolide/norethindrone in the treatment of endometriosis-associated chronic pelvic pain. This comparison will be based on a randomized, double-blind, trial of women with chronic pelvic pain who have been diagnosed with endometriosis at the time of surgery within the last 3 years. We hypothesize that, over a 12-month period of postoperative treatment, the efficacy of oral contraceptives is no worse than leuprolide/norethindrone, and that treatment with oral contraceptives is more cost-effective.

DETAILED DESCRIPTION:
* Background-Laparoscopic surgical treatment for endometriosis is typically associated with a decrease of pain on a short-term basis, but 50% of patients have pain 12 months after surgery. Often this leads to having repeat surgery to treat the endometriosis. Instead of having repeat surgery, some physicians use medications to prevent the pain and endometriosis from returning.
* The purpose of this study is to compare continuous oral contraceptives to depot-leuprolide for control of endometriosis-associated pelvic pain after surgical treatment of endometriosis. We will also be looking at the potential cost savings of using oral contraceptives compared to depot-leuprolide, as depot-leuprolide is an expensive medication.
* If the patient meets criteria, including confirmation of diagnosis of endometriosis, she will then undergo an intake visit consisting of obtaining informed consent and completion of several baseline questionnaires. This intake visit is estimated to last 1-2 hours. After informed consent has been obtained, the subject will be randomized to one of the two treatment groups:One tablet of oral contraceptives (birth control pills) everyday and an injection of saline (a sterile salt solution with no medication effect) every 12 weeks for 48 weeks or One tablet of norethindrone everyday and an injection of depot-leuprolide every 12 weeks for 48 weeks.
* The patient will be seen one month after the first injection (Visit 1) and then at 12 (Visit 2), 24 (Visit 3), 36 (Visit 4) and 48 (Visit 5) weeks. Blood pressure and weight will be recorded and a urine pregnancy test will be obtained. The Study Coordinator will review with the patient any concerns she might have and record any adverse events. Assessments of pain and quality of life will be made at weeks 4, 12, 24, 36 and 48 after the intake visit. An injection (leuprolide acetate or saline plus inert powder) will be given by an unblinded nurse at the intake visit, and at weeks 12, 24, and 36. In addition, at the end of each medication visit, the patient will be given a three month's supply of oral medication (capsules containing norethindrone acetate or a generic oral contraceptive with 30ug ethinyl estradiol and 0.15mg levonorgestrel).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 and pre-menopausal.
* Pelvic pain of at least 3 months duration.
* Diagnosis of endometriosis by laparoscopy or laparotomy within three years of entry. The diagnosis of endometriosis will require either histology consistent with endometriosis or operative records indicating visual evidence of lesions consistent with endometriosis.
* Moderate to severe pelvic pain preoperatively attributable to endometriosis (average Numerical Rating Scale of 5 or more for three or more months).
* Willingness to comply with visit schedule and protocol.

Exclusion Criteria:

* Use of oral contraceptives within one month of the surgery.
* Dose of Lupron within three months if given monthly or within five months if given 3-month injection.
* Any disorder that represents a contraindication to the use of oral contraceptives (e.g. insulin-dependent diabetes mellitus, history of thrombophlebitis, hypertension, history of cardiovascular disease, smoker at 35 or more years of age) or GnRH analogs (e.g., history of osteopenia).
* History of hysterectomy and bilateral salpingoophorectomy.
* Positive pregnancy test at first postoperative (i.e, intake visit).
* Significant mental or chronic systemic illness that might confound pain assessment or the inability to complete the study.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 194 (Estimated)
Dates: Start 2004-07

PRIMARY OUTCOMES:
pain
quality of life

CONTACTS AND LOCATIONS:
Overall Officials: David S Guzick, M.D., Ph.D, Principal Investigator — University of Rochester; Mark Hornstein, MD, Principal Investigator — Brigham and Women's Hospital; Fred M Howard, MD, Principal Investigator — University of Rochester; Sara Sukalich, MD, Principal Investigator — University of Rochester
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States